CLINICAL TRIAL: NCT04498299
Title: Stress Echocardiography in Patients Recovery From Mild COVID-19 Illness
Acronym: ECHO-vid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Miguel Ayala León (Network)
Responsible Party: Sponsor-Investigator, Miguel Ayala León, cardiovascular critical care unit director, Hospital Beneficencia Espanola de Puebla
Organization: Hospital Beneficencia Espanola de Puebla (Network)
Other Study IDs: Cardiology-004
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Echocardiography, Stress; COVID-19; Hypertension, Pulmonary
Keywords: Echocardiography, Stress; COVID-19; Pulmonary Hypertension
MeSH Terms: conditions — COVID-19; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: echocardiogram 2D — The patient is accelerating against a workload that gradually increases at a constant rate during the exercise, images will be obtained by echocardiography. The patient begins with 25 Watts with increments of 25 Watts every 3 minutes, continuing the exercise until significant electrocardiographic changes occur or the patient starts with symptoms.

SUMMARY:
With the appearance of the new SARS-COV2 virus, additional challenges are being imposed on the medical community after the resolution of acute COVID-19 illness, resulting in specific pathophysiologic mechanisms that while acutely damage the lung parenchyma might chronically impact the cardiopulmonary system.

This study aims to investigate changes after mild COVID-19 illness in echocardiographic indices at rest and stress.

ELIGIBILITY:
Inclusion Criteria:

* Having suffered mild COVID-19 illness
* PCR test negative after COVID-19 illness
* Men or women
* Age ≥18 years and < 45.
* No history of other cardiovascular or lung disease.
* No cardiovascular risk factors, that is, arterial systemic hypertension, smoking, diabetes, dyslipidemia
* No ongoing or previous cardio or vasoactive treatment
* Able to use the semi-supine exercise bicycle
* Able to give informed consent

Exclusion Criteria:

* Poor acoustic window.
* Tricuspid regurgitation more than mild
* Professional sports activity
* Pregnancy
* Obesity (body mass index [BMI], ≥30 kg/m2).
* Inability to provide consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients after the resolution of acute COVID-19 illness
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
• LA volume index | 3 minutes
  Left atrium volume index
• LV telediastolic diameter | 3 minutes
  Left ventricle telediastolic diameter
• LV telesystolic diameter | 3 minutes
  Left ventricle telesystolic diameter
• LV posterior wall | 3 minutes
  Left ventricle posterior wall
• RA area | 3 minutes
  Right atrium area
• RV basal dimensión | 3 minutes
  Right ventricle basal dimensión
• RV mid cavity dimension; | 3 minutes
  Right ventricle cavity dimensión
• RV longitudinal dimension | 3 minutes
  Right ventricle longitudinal dimension
• Distal, RV outflow tract dimension at the distal or pulmonic valve level | 3 minutes
  Distal, right ventricle outflow tract dimension at the distal or pulmonic valve level
• Proximal RV outflow tract dimension at the proximal subvalvular level | 3 minutes
  Proximal right ventricle outflow tract dimension at the proximal subvalvular level
• TAPSE | 3 minutes
  • Tricuspid annular plane systolic excursion
• RV free Wall strain | 3 minutes
  Right ventricle free Wall strain
• Inferior cava vein PW Doppler | 3 minutes
  Inferior cava vein PW Doppler
• E wave mitral | 3 minutes
  E wave mitral
• A wave mitral | 3 minutes
  A wave mitral
• E wave /A wave mitral | 3 minutes
  E wave /A wave mitral
• E-wave at mitral annulus | 3 minutes
  E-wave at mitral annulus
• E-wave at mitral annulus / A-wave at the mitral annulus | 3 minutes
  E-wave at mitral annulus / A-wave at the mitral annulus
• E wave/ E-wave at the mitral annulus | 3 minutes
  E wave/ E-wave at the mitral annulus
• E tricuspid (E) | 3 minutes
  E tricuspid (E)
• A tricuspid (A) | 3 minutes
  A triuspid (A)
• E/A | 3 minutes
  E/A
• Systolic pulmonary artery pressure | 3 minutes
  Systolic pulmonary artery pressure
• E-wave at the tricuspid annulus | 3 minutes
  E-wave at the tricuspid annulus
• Mean pulmonary artery pressure | 3 minutes
  Mean pulmonary artery pressure
• Stroke volume | 3 minutes
  Stroke volume
• Cardiac output | 3 minutes
  Cardiac output

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Beneficencia Española de Puebla, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No